CLINICAL TRIAL: NCT06248736
Title: Description of Lactulose Administration by Balloon Rectal Tube in Severe Hepatic Encephalopathy
Acronym: ALPACA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: CHU Grenoble/ ALPACA
Record Dates: First submitted 2023-11-14; First posted 2024-02-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Acute liver failure in cirrhotic patients is associated with a one-month mortality of 48%. Encephalopathy, largely related to hyperammonemia, is a frequent complication of liver failure and is a poor prognostic marker. Lactulose decreases ammonia by acidification of the colon, replacement of urease-producing bacteria and creation of a laxative effect. Thus, the administration of lactulose in patients with severe hepatic encephalopathy reduces mortality by more than 40%.

In intensive care patients, lactulose is often administered rectally. The use of simple rectal tubes is associated with frequent leakage of lactulose as well as faecal discharge and therefore risks of infection and skin lesions. Balloon rectal tubes with a drug delivery valve have recently been developed and used in this indication. The aim of this study is therefore to describe the use of these balloon rectal tubes to administer Lactulose in severe hepatic encephalopathy.

This suggests that ammonia reduction in these patients may prolong survival time.

No studies have described the administration of Lactulose via the rectal route with a balloon tube. The descriptive methodology is therefore appropriate. This is a preliminary study allowing data collection to establish the methodology for a subsequent clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Patients treated with Lactulose with balloon rectal probe

Exclusion Criteria:

* Patient(s) objecting to the use of their data for research purposes
* Rectal probe contraindication: damage to the rectal mucosa, rectal surgery, severe haemorrhoids, rectal stenosis, rectal tumour,
* Lactulose contraindication (person unable to absorb galactose)
* Patients deprived of liberty, under guardianship or curators
* Pregnant women
* Patient not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe hepatic encephalopathy hospitalised in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Describe ammonia during lactulose administration by balloon rectal tube | 48 hours
  Variation of ammonia before treatment and after 48h of treatment

SECONDARY OUTCOMES:
Describe the neurological course following administration of lactulose via a balloon rectal tube | at 7 days
  Score Richmond Agitation-Sedation Scale from the minimum value -4 to maximum value + 4 Richmond Agitation and sedation scale , agitation
Describe ammonia levels after lactulose administration via balloon rectal tube. | at 7 days
  Change in ammonia over 1 week in µmol/l after administration
Describe the skin tolerance of patients during hospitalization. | at 7 days
  Percentage of patients with at least one pressure sore or infection in the lumbar, pelvic, buttocks, or buttock area
Describe complications related to the balloon rectal tube | at 7 days
  Percentage of patients with at least one of the following complications: leakage of faeces during or after use of the catheter; rectal bleeding; peri-anal skin damage (fissure, ulcer, infection); bowel obstruction; bowel perforation, rectal pain, abdominal distension.
Describe complications related to rectal lactulose administration | at 7 days
  Percentage of patients with at least one of the following complications: hypernatremia > 150 mmol/L, dehydration, renal insufficiency urea creatinemia.
Patient outcomes | at 28 days
  Duration of invasive ventilation, duration of resuscitation or intensive care, duration of hospital stay, mortality
Caregiver satisfaction | at 7 days
  Anonymised use and maintenance satisfaction questionnaire into 0 is the worst score and 10 is the better score
Describe balloon rectal probe retention | at 7 days
  Frequency of leakage during and within one hour of lactulose administration when the rectal probe balloon is inflated

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUZAT, recruting, Principal Investigator — CENTRE HOSPITALIER UNIVERSITAIRE GRENOBLE ALPES
Locations (1):
- Pr PIERRE BOUZAT, Grenoble, France

REFERENCES:
- [Background] Clemmesen JO, Larsen FS, Kondrup J, Hansen BA, Ott P. Cerebral herniation in patients with acute liver failure is correlated with arterial ammonia concentration. Hepatology. 1999 Mar;29(3):648-53. doi: 10.1002/hep.510290309. PMID 10051463
- [Background] Shalimar, Sheikh MF, Mookerjee RP, Agarwal B, Acharya SK, Jalan R. Prognostic Role of Ammonia in Patients With Cirrhosis. Hepatology. 2019 Sep;70(3):982-994. doi: 10.1002/hep.30534. Epub 2019 Mar 21. PMID 30703853
- [Background] Dasarathy S, Mookerjee RP, Rackayova V, Rangroo Thrane V, Vairappan B, Ott P, Rose CF. Ammonia toxicity: from head to toe? Metab Brain Dis. 2017 Apr;32(2):529-538. doi: 10.1007/s11011-016-9938-3. Epub 2016 Dec 24. PMID 28012068
- [Background] Jalan R, De Chiara F, Balasubramaniyan V, Andreola F, Khetan V, Malago M, Pinzani M, Mookerjee RP, Rombouts K. Ammonia produces pathological changes in human hepatic stellate cells and is a target for therapy of portal hypertension. J Hepatol. 2016 Apr;64(4):823-33. doi: 10.1016/j.jhep.2015.11.019. Epub 2015 Dec 2. PMID 26654994
- [Background] Ravi S, Bade KS, Hasanin M, Singal AK. Ammonia level at admission predicts in-hospital mortality for patients with alcoholic hepatitis. Gastroenterol Rep (Oxf). 2017 Aug;5(3):232-236. doi: 10.1093/gastro/gow010. Epub 2016 May 1. PMID 27132633
- [Background] Bhatia V, Singh R, Acharya SK. Predictive value of arterial ammonia for complications and outcome in acute liver failure. Gut. 2006 Jan;55(1):98-104. doi: 10.1136/gut.2004.061754. Epub 2005 Jul 15. PMID 16024550
- [Background] Bernal W, Hall C, Karvellas CJ, Auzinger G, Sizer E, Wendon J. Arterial ammonia and clinical risk factors for encephalopathy and intracranial hypertension in acute liver failure. Hepatology. 2007 Dec;46(6):1844-52. doi: 10.1002/hep.21838. PMID 17685471